CLINICAL TRIAL: NCT04208841
Title: Strengthening Person-centered Accessibility, Respect, and Quality of Maternal Health Services in India, Phase 2
Brief Title: Quality Improvement of Person-Centered Care for Maternal Health in Public Facilities in India, Phase 2
Acronym: SPARQINDIA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Population Services International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-18008_QI India_Phase2
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Reproductive Health
Keywords: Maternal Health; India; Person-Centered Care; Quality Improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control - Patient (No Intervention): Participants who receive maternal health services at a facility not participating in the Quality Improvement Intervention or implementing the change package
- Sustaining - Patients (Experimental): Participants who received maternal health services at a facility where a quality improvement collaborative had been implemented
  Interventions: Behavioral: Person-Centered Care Quality Improvement Collaborative Sustain
- Spread - Patients (Experimental): Participants who received maternal health services at a facility that was provided a change package of ideas developed during the quality improvement collaborative (in phase 1) and used to make improvements on person-centered care
  Interventions: Behavioral: Person-Centered Care Quality Improvement Collaborative Spread
- Control - Providers (No Intervention): Providers who work at a facility not participating in the Quality Improvement Intervention or implementing the change package
- Sustaining - Providers (Experimental): Providers who work at a facility where a quality improvement collaborative had been implemented
  Interventions: Behavioral: Person-Centered Care Quality Improvement Collaborative Sustain
- Spread - Providers (Experimental): Participants who work at a facility that was provided a change package of ideas developed during the quality improvement collaborative (in phase 1) and used to make improvements on person-centered care
  Interventions: Behavioral: Person-Centered Care Quality Improvement Collaborative Spread

INTERVENTIONS:
Behavioral: Person-Centered Care Quality Improvement Collaborative Sustain — Sustain improvements during QI collaborative focused on PCC
  Arms: Sustaining - Patients; Sustaining - Providers
Behavioral: Person-Centered Care Quality Improvement Collaborative Spread — Implement change package developed during QI Collaborative
  Arms: Spread - Patients; Spread - Providers

SUMMARY:
Evaluating the spread of a quality improvement (QI) change package working to improve person-centered care (PCC) for maternal health (MH) services.

DETAILED DESCRIPTION:
After implementing a quality improvement (QI) collaborative in public facilities in Uttar Pradesh, India, a second phase was done to evaluate if the "change package" developed during phase one could be implemented in similar facilities to improve the quality of person-centered care (PCC) for a maternal health (MH) services.

ELIGIBILITY:
Inclusion Criteria for Women:

* Women aged 18-49 years old
* Who agreed to participate
* Who delivered a baby at the facility where data collection is taking place within the last 7 days

Exclusion Criteria for Women:

* Not a women aged 18-49
* Did not agree to participate
* Did not deliver a baby at the facility where data collection is taking place within the last 7 days

Inclusion Criteria for Providers:

* Agreed to participate
* Purposive sampling
* Permanent staff at the facility

Exclusion Criteria for Providers:

* Did not agree to participate
* Not permanent staff at the facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1971 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Person-Centered Maternal Health Scale Score | baseline
  Survey conducted with women: self-report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person-Centered Maternal Health Scale Score | About 12 month post baseline
  Survey conducted with women: self-report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person-Centered Scale Score | baseline
  Survey conducted with providers: self-report of perceptions of care. Possible range 0-100; higher the score the better the experience of care
Person-Centered Scale Score | About 12 months post baseline
  Survey conducted with providers: self-report of perceptions of care. Possible range 0-100; higher the score the better the experience of care

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Monatgu, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Population Services International, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sudhinaraset M, Giessler K, Nakphong MK, Roy KP, Sahu AB, Sharma K, Montagu D, Green C. Can changes to improve person-centred maternity care be spread across public health facilities in Uttar Pradesh, India? Sex Reprod Health Matters. 2021 Dec;29(1):1-15. doi: 10.1080/26410397.2021.1892570. PMID 33704027
- [Derived] Montagu D, Giessler K, Nakphong MK, Green C, Roy KP, Sahu AB, Sharma K, Sudhinarset M. A comparison of intensive vs. light-touch quality improvement interventions for maternal health in Uttar Pradesh, India. BMC Health Serv Res. 2020 Dec 4;20(1):1121. doi: 10.1186/s12913-020-05960-6. PMID 33276773